CLINICAL TRIAL: NCT02585544
Title: Ambulatory Prolapse Surgery: Feasibility Study
Brief Title: Ambulatory Prolapse Surgery
Acronym: PROLAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL15_0215; 2015-A00599-40 (Other: ID-RCB)
Record Dates: First submitted 2015-10-19; First posted 2015-10-23 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Genital Prolapse; Vaginal Floor Prolapse
Keywords: genital prolapse; day-care management; vaginal route; prosthetic reinforcement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genital prolapse (Other): Single arm: i.e., all patients
  Interventions: Procedure: day-care surgery

INTERVENTIONS:
Procedure: day-care surgery — day-care surgery

SUMMARY:
Day surgery is performed in the same way as in full hospital admission, allowing same-day discharge without increased risk. It provides many grounds for patient satisfaction. Progress in surgical and anesthesia techniques now allows this form of management to be developed and prioritized.

Day-care surgery for prolapse has been little studied. The present study is intended to help extend its future implementation, the primary objective being to assess the feasibility of the day-care approach in prolapse surgery. The secondary objectives are to study criteria of non-eligibility for day-care prolapse surgery, reasons for patients' refusal, causes of failure, predictive factors for failure, patient satisfaction, postoperative complications, 2-year anatomic and functional results, pain, quality of life and sexuality, and postoperative onset of dyspareunia and urinary incontinence.

The design is for a prospective non-randomized study conducted in 3 gynecologic surgery sites managed by the Lyon hospitals board (Hospices Civils de Lyon).

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV anterior genital prolapse (cystocele) on the Pelvic Organ Prolapse Quantification (POP-Q) classification and/or vaginal floor prolapse
* Vaginal approach with prosthetic reinforcement planned
* Patient eligible for day-surgery
* Patient consenting to participate
* Informed and signed consent

Exclusion Criteria:

* Interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, progressive disease, etc.
* Patient with ≥1 ineligibility criterion for day-surgery
* Impaired lower-limb range of motion preventing positioning for surgery
* Pregnancy, ongoing or planned during the study period
* Progressive or latent infection or signs of tissue necrosis on clinical examination
* Non-controlled diabetes (glycated hemoglobin >8%)
* Treatment impacting immune response (immunomodulators), ongoing or within previous month
* History of pelvic region radiation therapy, at any time
* History of pelvic cancer
* Non-controlled progressive spinal pathology
* Known hypersensitivity to one of the implant components (polypropylene)
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Number of patient with success for ambulatory surgery | Day 1 (postoperative)
  Number of prolapse surgery patients actually managed on a day-care basis

SECONDARY OUTCOMES:
causes of non-eligibility for day-care management analysis | Day 1 (before surgery)
  list and percentage
reasons for patients' refusal analysis | Day 1 (before surgery)
  list and percentage
causes of failure of day-surgery analysis | Day 1 (postoperative)
  list and percentage
Number of patients satisfied with day-surgery | Day 1 (postoperative)
Post-surgery complications | Day 1 (postoperative), month 1, year 1 and year 2
  number and percentage of cases of infection, hematoma, urinary retention, healing defect (exposure or erosion), retraction, death
Number of prolapse correction failure | month 1, year 1 and year 2
pain score analysis | month 1, year 1 and year 2
  0 to 10 scale
quality of life scores analysis | month 1, year 1 and year 2
  SF- 12 Short Form (12) Health Survey PFDI-20 : Pelvic Floor Distress Inventory PFIQ-7 : Pelvic Floor Impact Questionnaire PGI-I : Patient Global Impression of Improvement
quality of life scores analysis | month 1, year 1 and year 2
  SF- 12 Short Form (12) Health Survey
quality of life scores analysis | month 1, year 1 and year 2
  PFDI-20 : Pelvic Floor Distress Inventory
quality of life scores analysis | month 1, year 1 and year 2
  PGI-I : Patient Global Impression of Improvement
quality of life scores analysis | month 1, year 1 and year 2
  PFIQ-7 : Pelvic Floor Impact Questionnaire
sexuality score analysis | month 1, year 1 and year 2
  PISQ-12 questionnaire
percentage dyspareunia | month 1, year 1 and year 2
number of onset of urinary incontinence | month 1, year 1 and year 2

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

REFERENCES:
- [Background] Lamblin G, Courtieu C, Bensouda-Miguet C, Panel L, Moret S, Chabert P, Chene G, Nohuz E. Outpatient vaginal surgery for pelvic organ prolapse: a prospective feasibility study. Minerva Ginecol. 2020 Feb;72(1):19-24. doi: 10.23736/S0026-4784.20.04510-4. PMID 32153159